CLINICAL TRIAL: NCT06647940
Title: Orelabrutinib in Combination with R-CHOP for CD5-positive DLBCL Patients: a Single-arm, Multicenter, Phase II Clinical Trial（Rocket Trial）
Brief Title: Orelabrutinib in Combination with R-CHOP for CD5-positive DLBCL Patients（Rocket Trial）
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Fifth Affiliated Hospital, Sun Yat-Sen University (Other); Gansu Cancer Hospital (Other); First Affiliated Hospital of Shantou University Medical College (Other); Southern Medical University, China (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Fifth Affiliated Hospital of Guangzhou Medical University (Other); Shenzhen People's Hospital (Other); Guangzhou First People's Hospital (Other); Dongguan People's Hospital (Other Government); The First People's Hospital of Zhaoqing (Unknown)
Responsible Party: Principal Investigator, Qingqing Cai, chief physician, Sun Yat-sen University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2024-570-01
Record Dates: First submitted 2024-10-16; First posted 2024-10-18 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Diffuse Large B Cell Lymphoma (DLBCL)
Keywords: DLBCL; Orelabrutinib; CD5-positive; R-CHOP
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — orelabrutinib; R-CHOP protocol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Orelabrutinib in combination with R-CHOP (Experimental): Patients with CD5 positive diffuse large B-cell lymphoma will receive orelabrutinib in combination with R-CHOP regimen from the second cycle of R-CHOP (3 weeks per cycle).
  After 8 cycles of induction therapy, if the response is assessed as complete remission (CR), maintenance therapy with orelabrutinib will be conducted.
  Interventions: Drug: Orelabrutinib Oral Tablet; Drug: R-CHOP Protocol

INTERVENTIONS:
Drug: Orelabrutinib Oral Tablet — Orelabrutinib (150 mg po D1-D21) is added from the second cycle of R-CHOP regimen
  Other Names: Bruton's Tyrosine Kinase Inhibitor
Drug: R-CHOP Protocol — Rituximab, Cyclophosphamide, Doxorubicin, Vincristine, Prednisone
  Other Names: R-CHOP regimen

SUMMARY:
This is a prospective, single-arm, multicenter, phase II clinical trial to evaluate the efficacy and safety of orelabrutinib combined with the R-CHOP (rituximab, cyclophosphamide, vincristine, doxorubicin, and prednisone) regimen as first-line treatment in CD5-positive diffuse large B-cell lymphoma (DLBCL) patients.

DETAILED DESCRIPTION:
The purpose of this phase II clinical trial is to evaluate the efficacy and safety of orelabrutinib in combination with R-CHOP for untreated CD5-positive DLBCL patients.

The induction phase consisted of 6 cycles of orelabrutinib in combination with R-CHOP (orelabrutinib added from the second cycle), followed by 2 cycles of rituximab + orelabrutinib, for a total of 8 treatment cycles. After 8 cycles of induction therapy, if the response is assessed as complete remission (CR), maintenance therapy with orelabrutinib will be conducted.

The primary endpoint is the 2-year event-free survival (EFS) rate.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign informed consent.
2. Aged ≥18 years, both male and female.
3. Pathologically confirmed CD5-positive DLBCL
4. There must be at least one measurable or evaluable lesion that meets the evaluation criteria for Lugano 2014 lymphoma.
5. Eastern Cooperative Oncology Group(ECOG) performance status score of 0-2.
6. Expected survival ≥3 months.
7. Sufficient bone marrow, liver, and kidney function.

Key Exclusion Criteria:

1. DLBCL combined with other types of lymphoma. Transformed DLBCL.
2. DLBCL with central nervous system invasion.
3. The patients had previously received BTK inhibitors.
4. The patients have contraindications to any drug in the combined treatment.
5. Patients with the infection of human immunodeficiency virus (HIV) and/or acquired immunodeficiency syndrome.
6. Inability to swallow tablets, presence of malabsorption syndrome, or any other gastrointestinal disease or dysfunction that may affect the absorption of the study drug.
7. Pregnant and lactating women, and subjects of childbearing age who do not want to use contraception.
8. Mentally ill persons or persons unable to obtain informed consent.
9. The investigators think that the patient is not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-11-01 (Estimated); Primary Completion 2026-11-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
2-year event-free survival (EFS) rate | Defined as the proportion of patients without disease progression, treatment discontinuation, or death for any reason within 24 months of enrollment
  To investigate the preliminary anti-tumor efficacy

SECONDARY OUTCOMES:
Complete response rate (CRR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy
Disease-free survival (DFS) | From date of the first complete response until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Objective response rate (ORR) | Up to 8 cycles (each cycle is 21 days)
  To investigate the preliminary anti-tumor efficacy
Progression-free survival (PFS) | From the date of enrollment until the date of the first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Overall survival (OS) | From the date of enrollment until the date of death from ant cause, assessed up to 24 months
  To investigate the preliminary anti-tumor efficacy
Number of participants with adverse events (AE) and severe adverse events (SAE) as assessed by CTCAE v5.0 | Through study completion, an average of 2 years
  To identify the incidence of AE and SAE

OTHER OUTCOMES:
The correlation of gene mutations and alterations in relevant signaling pathways with the efficacy and survival in CD5-positive DLBCL | Through study completion, an average of 2 years
  To explore the correlations between gene mutations and response and prognosis

CONTACTS AND LOCATIONS:
Locations (11):
- China (11):
  - Sun Yat-sen Universitiy Cancer Center, Sun Yat-Sen University,, Guangzhou, China
  - Gansu Cancer Hospital, Lanzhou, Gansu
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Fifth Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First People's Hospital of Guangzhou, Guangzhou, Guangdong
  - Guangdong Provincial Hospital of Traditional Chinese Medicine, Guangzhou, Guangdong
  - Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - First Affiliated Hospital of Shantou University Medical College., Shantou, Guangdong
  - Shenzhen People's Hospital, Shenzhen, Guangdong
  - Zhaoqing First People's Hospital, Zhaoqing, Guangdong
  - Fifth Affiliated Hospital of Sun Yat-sen University, Zhuhai, Guangdong

IPD SHARING:
Plan to Share IPD: Undecided